CLINICAL TRIAL: NCT02404753
Title: A Randomized, Single Center, Controlled Phase II Study to Compare Laparoscopic Versus Open Distal Gastrectomy in Locally Advanced Gastric Cancer After Neoadjuvant Chemotherapy
Brief Title: A Comparison of Laparoscopic With Open Distal Gastrectomy in Advanced Gastric Cancer After Neoadjuvant Chemotherapy
Acronym: REALIZATION
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Ziyu Li, MD, Chief Physician,Associate Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GISCA2015001/LAP
Record Dates: First submitted 2015-03-23; First posted 2015-03-31 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Gastric Cancer
Keywords: Locally advanced gastric cancer; Laparoscopic distal D2 gastrectomy; Neoadjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic gastrectomy (Experimental): Laparoscopic distal gastrectomy and D2 lymph node dissection are performed for locally advanced gastric cancer after neoadjuvant chemotherapy.
  Interventions: Drug: Neoadjuvant Chemotherapy; Procedure: Laparoscopic gastrectomy; Drug: Adjuvant Chemotherapy
- Open gastrectomy (Active Comparator): Open distal gastrectomy and D2 lymph node dissection are performed for locally advanced gastric cancer after neoadjuvant chemotherapy.
  Interventions: Drug: Neoadjuvant Chemotherapy; Procedure: Open gastrectomy; Drug: Adjuvant Chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy — XELOX: Oxaliplatin 130mg/m2,iv.,d1;Capecitabine 1000mg/m2,po.,Bid,d1-14; Repeat every 21 days for 3 courses.
  Other Names: NACT
Procedure: Laparoscopic gastrectomy — Laparoscopic distal gastrectomy with D2 lymph node dissection
  Other Names: LDG
  Arms: Laparoscopic gastrectomy
Procedure: Open gastrectomy — Open distal gastrectomy with D2 lymph node dissection
  Other Names: ODG
  Arms: Open gastrectomy
Drug: Adjuvant Chemotherapy — XELOX: Oxaliplatin 130mg/m2,iv.,d1;Capecitabine 1000mg/m2,po.,Bid,d1-14; Repeat every 21 days for 5 courses.
  Other Names: ACT

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of laparoscopic distal D2 gastrectomy (LDG) compared with open surgery (ODG) for resectable gastric cancer, to determine whether LDG can be a test arm for a future Phase III trial to evaluate the non-inferiority of overall survival compared with ODG in patients who receive neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
The study is an open-label, controlled, randomized Phase II clinical trial. The protocol has been approved by the Ethics Committee of Beijing Cancer Hospital.

The primary endpoint is the 3-year progression-free survival (PFS) rate. The secondary endpoints are the overall survival, surgical morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the stomach.
* Clinical cT2N+M0,or cT3-4a/N+M0 disease, confirmed by upper gastrointestinal endoscopy and abdominal computed tomography (CT) and laparoscopy. The T and N stages are determined by the method of Habermann et al.
* The gastric tumors are located in the middle to lower third of the stomach, are macroscopically resectable by distal gastrectomy with D2 lymph node dissection, and R0 or R1 resection can be achieved.
* No bulky lymph node metastasis is detected by abdominal CT.
* No pleural effusion, no ascites exceeding the pelvis and no metastasis to the peritoneum, liver or other distant organs are confirmed by abdominal pelvic CT.
* No clinically apparent distant metastasis.
* Karnofsky performance status ≥70%.
* Sufficient oral intake.
* No previous treatment with chemotherapy or radiation therapy for any tumors.
* No previous surgery for the present disease.
* Sufficient organ function, as evaluated by laboratory tests 7 days or more after the date when the anticancer drugs were given. When patients are recovering from myelosuppression,the revised criteria are shown in parentheses.

White blood cell count≥3000/mm3 (2000/mm3) Platelet count≥10.0*104/mm3 (5.0*104/mm3) Aspartate aminotransferase≤100 IU/l Alanine aminotransferase≤100 IU/l Total bilirubin≤2.0 mg/dl Serum creatinine≤1.5 mg/dl

* No need for emergency surgery due to bleeding or perforation of the primary tumor.
* No mechanical obstruction.
* Written informed consent.

Exclusion Criteria:

* Past history of upper abdominal surgery.
* Past history of surgery for the gastrointestinal tract.
* Body mass index exceeding 30 kg/m2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-11-25 (Estimated); Study Completion 2022-11-25 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival | 36 months
  In terms of locally advanced gastric cancer, to evaluate the disease free survival rate in laparoscopic subtotal gastrectomy with D2 lymph node dissection at postoperative 3 years compared with open subtotal gastrectomy with D2 lymph node dissection

SECONDARY OUTCOMES:
Overall survival | 36 months
  In terms of locally advanced gastric cancer, to evaluate the overall survival rate in laparoscopic subtotal gastrectomy with D2 lymph node dissection at postoperative 3 years compared with open subtotal gastrectomy with D2 lymph node dissection
Surgical morbidity | 30 days
  Surgical morbidity is defined as the events which occurs with-in postoperative 30 days, extension of hospitalization and re-hospitalization. It is necessary to evaluate the complication and if it occurs during the hospitalization, it is required to record complication name, date of on-set (postoperatively), grade on Clavien-Dindo Classification and treatment for complication.
Surgical mortality | 30 days
  It is defined as the death within postoperative 30 days regardless of postoperative reason. If the patient is transferred to other medication institutes with impossible condition for recovery before death, it is regarded as death.
Postoperative recovery index | 2 weeks
  Postoperatively, the investigator evaluates the patient's recovery condition once a day. Evaluation items for patient's recovery condition: the pain score, the leaving bed time, postoperative gastrointestinal function recovery time and hospital stay.
Postoperative quality of life | Up to 1 year post-operative
  In pre-therapy <7 days, pre-operative <7 days, and post-operative at 12 months after surgery, both the European Organisation for Research and Treatment of Cancer (EORTC) C30 and STO22 are analyzed with quality of life by following methods. In case of EORTC-C30, the analysis is undergone by classifying into 5 functional scales (physical, role, emotional, cognitive, and social functioning), 3 symptom scales (fatigue, pain and nausea, and vomiting), 1 global health status and 6 single items.

CONTACTS AND LOCATIONS:
Overall Officials: Ziyu Li, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Li Z, Shan F, Ying X, Zhang L, Ren H, Li S, Jia Y, Miao R, Xue K, Li Z, Wang Y, Yan C, Zhang Y, Pang F, Ji J. Laparoscopic or open distal gastrectomy after neoadjuvant chemotherapy for advanced gastric cancer: study protocol for a randomised phase II trial. BMJ Open. 2018 Aug 10;8(8):e021633. doi: 10.1136/bmjopen-2018-021633. PMID 30099396
- [Background] Li Z, Shan F, Wang Y, Li S, Jia Y, Zhang L, Yin D, Ji J. Laparoscopic versus open distal gastrectomy for locally advanced gastric cancer after neoadjuvant chemotherapy: safety and short-term oncologic results. Surg Endosc. 2016 Oct;30(10):4265-71. doi: 10.1007/s00464-015-4739-z. Epub 2016 Jun 10. PMID 27287914
- [Derived] Li Z, Shan F, Ying X, Zhang Y, E JY, Wang Y, Ren H, Su X, Ji J. Assessment of Laparoscopic Distal Gastrectomy After Neoadjuvant Chemotherapy for Locally Advanced Gastric Cancer: A Randomized Clinical Trial. JAMA Surg. 2019 Dec 1;154(12):1093-1101. doi: 10.1001/jamasurg.2019.3473. PMID 31553463

DOCUMENTS (2):
  • Study Protocol (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT02404753/Prot_000.pdf
  • Informed Consent Form (2015-02-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT02404753/ICF_001.pdf